CLINICAL TRIAL: NCT03178357
Title: "Efficacy and Safety of Cardiac Rehabilitation in Patients With Hypertrophic Cardiomyopathy Without Left Ventricular Outflow Tract Obstruction With Preserved Systolic Function - Pilot Study".
Brief Title: "Cardiac Rehabilitation in Patients With Hypertrophic Cardiomyopathy".
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2.1/I/17
Record Dates: First submitted 2017-06-05; First posted 2017-06-06 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Cardiac Rehabilitation
MeSH Terms: interventions — Cardiac Rehabilitation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCM patients with CR (Other): 30 HCM patients treated as standard subjected to 4-week hospital cardiac rehabilitation (CR) including psychological care (counseling and / or psychoeducation) and physical training followed by 8 weeks of telerehabilitation in the patient's home (cardiac rehabilitation + standard therapy)
  Interventions: Other: Cardiac rehabilitation + standard therapy
- HCM patients without CR (control group) (Other): 30 HCM patients in control group - standard treatment according to current guidelines and outpatient visits with psychological and / or psychoeducational counseling (standard therapy)
  Interventions: Other: Standard therapy

INTERVENTIONS:
Other: Cardiac rehabilitation + standard therapy — Patients with HCM subjected to cardiological rehabilitation
  Other Names: Standard therapy
  Arms: HCM patients with CR
Other: Standard therapy — Standard treatment according to current guidelines and outpatient visits with psychological and / or psychoeducational counseling
  Arms: HCM patients without CR (control group)

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is the most common hereditary disease characterized by left ventricular hypertrophy and consequently left ventricular diastolic dysfunction. Its prevalence is estimated at around 0.2% in the general population. HCM is the most common cause of sudden cardiac death due to cardiovascular disease in young athletes, accounting for one third of deaths. HCM patients often have symptoms of heart failure. The ESC recommendations for heart failure (HF) from 2016 recommend exercise training regardless of ejection fraction to improve exercise capacity, quality of life, and reduction in hospitalizations due to HF. Meanwhile, for many years, HCM was equivalent to exercise training limitation. According to the 2014 ESC guidelines, it is recommended for patients with HCM to avoid sports practice. However the results of Edelmann et al. research, suggest that physical training leads to a significant clinical improvement in patients with diastolic dysfunction and thus may be beneficial in patients with HCM. In 2015 results of a first study were published (Klempfner et al.), which showed that the majority of HCM patients with moderate risk undergoing supervised physical training had improved physical performance and no significant adverse events were recorded. The study was limited by the small number of admitted patients (twenty), lack of control group and failure to perform cardio-pulmonary exercise test.

The main goal of the study will be to evaluate the effectiveness and safety of comprehensive cardiological rehabilitation and telerehabilitation in patients with hypertrophic cardiomyopathy without left ventricular outflow tract obstruction with preserved systolic function. The study is planned to include 30 patients with HCM subjected to physical training and 30 patients with HCM in the control group treated as standard according to current guidelines, not subjected to physical training.

DETAILED DESCRIPTION:
The main goal of the study will be to evaluate the effectiveness and safety of comprehensive cardiological rehabilitation and telerehabilitation in patients with hypertrophic cardiomyopathy without left ventricular outflow tract obstruction with preserved systolic function. The study is planned to include 30 patients with HCM subjected to physical training and 30 patients with HCM in the control group treated as standard according to current guidelines, not subjected to physical training.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with hypertrophic cardiomyopathy (defined in accordance with the ESC guidelines for the diagnosis and management of cardiomyopathy and hypertrophy in 2014): thickness ≥ 15 mm of one or more segments of the left ventricular wall measured using any imaging technique [echocardiography, cardiac magnetic resonance or computed tomography] which can not be explained solely by the left ventricular loading conditions) without left ventricular outflow tract obstruction at rest: gradient <30 mmHg.
2. Stable general condition (1 month period).
3. NYHA Class II and III.
4. Preserved LV systolic function (LVEF ≥ 50%).
5. Condition after ICD implantation.
6. Written informed consent of the patient to participate in the Program.
7. Completed eighteen years of age.

Exclusion Criteria:

1. Complex life-threatening ventricular arrhythmias that can not be treated.
2. Uncontrolled hypertension.
3. Advanced atrio-ventricular block.
4. Myocarditis or pericarditis (up to 6 months).
5. Symptomatic aortic stenosis.
6. Acute systemic illness.
7. Intracardiac thrombosis.
8. Significant ischaemia during low intensity exercise test (2 METS, 50W).
9. Uncontrolled diabetes.
10. Pulmonary embolism (up to 6 months).
11. Thrombophlebitis.
12. New episode of AF/Afl.
13. Decrease in systolic blood pressure during exercise.
14. Co-morbidities that limit exercise tolerance and prevent exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 | 36 months
  Physical efficiency evaluated in the measurable parameter - peak VO2.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Sadowski, Principal Investigator — The Cardinal Stefan Wyszyński Institute of Cardiology
Locations (1):
- The Cardinal Stefan Wyszyński Institute of Cardiology, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No